CLINICAL TRIAL: NCT06490198
Title: A Single-Arm, Phase 2 Study to Evaluate OBI-833/OBI-821 Maintenance Therapy in Patients With Globo H-Positive Advanced Biliary Tract Cancer Not Progresseding Under First-Line Gemcitabine and Cisplatin
Brief Title: Phase 2 Study: OBI-833/OBI-821 Maintenance for Globo H+ Advanced Biliary Tract Cancer After Gemcitabine/Cisplatin
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yeh Chun-Nan, Professor and Chief Department of Surgery, Chang Gung Memorial Hospital, Linkou and Chang Gung University, Taipei, Taiwan, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202400601A0C601
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Cholangiocarcinoma; Chemotherapy Effect; Immunotherapy
Keywords: Cholangiocarcinoma; Immunotherapy; Chemotherapy; Globo-H
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Globo-H (Experimental): OBI-833, 30 μg/ OBI-821 100 μg, Subcutaneous injection at Weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 32, 40, 48, 56, 64, 72, and 80 weeks
  Interventions: Drug: OBI-833/OBI-821

INTERVENTIONS:
Drug: OBI-833/OBI-821 — OBI-833 is a glycoconjugate that consists of Globo H, a unique tumor-associated carbohydrate antigen (TACA), covalently linked to cross-reacting material 197 (CRM197), an inactive and nontoxic form of diphtheria toxin (DT) acting as the carrier protein.
  OBI-821 is a saponin-based adjuvant derived from the bark of the Quillaja saponaria Molina tree. It is a purified saponin adjuvant structurally similar to adjuvant QS-21. The OBI-833/OBI-821 combination represents a carbohydrate-conjugate vaccine combined with an immune adjuvant, intended to serve as an active cancer immunotherapy.
  Other Names: Globo H-CRM197

SUMMARY:
A Phase 2 clinical trial protocol for evaluating the efficacy and safety of OBI-833/OBI-821, a carbohydrate-conjugate vaccine combined with an immune adjuvant, as maintenance therapy in combination with first-line gemcitabine and cisplatin chemotherapy for patients with Globo H-positive advanced biliary tract cancer. The study is designed as a single-arm trial with 30 patients who have achieved stable disease, partial response, or complete response after 3±1 months of initial chemotherapy. The primary endpoint is progression-free survival, with secondary endpoints including overall survival, tumor response, and safety profile. The treatment regimen involves subcutaneous injections of OBI-833/OBI-821 on a gradually decreasing frequency schedule for up to 80 weeks. The trial also includes exploratory objectives to assess immune responses and biomarkers. This study aims to address the unmet need for improved treatment options in advanced biliary tract cancer by leveraging the potential of immunotherapy targeting the Globo H antigen.

DETAILED DESCRIPTION:
This clinical trial is a single-arm, phase 2 study evaluating OBI-833/OBI-821 as maintenance therapy in patients with Globo H-positive advanced biliary tract cancer who have not progressed on first-line gemcitabine and cisplatin chemotherapy. The study is grounded in the challenging prognosis of biliary tract cancer, including cholangiocarcinoma, which has limited treatment options. Currently, the standard first-line therapy is gemcitabine plus cisplatin, but progression-free survival remains short at around 6 months, highlighting the need for improved treatment strategies.

The investigational therapy, OBI-833, is a glycoconjugate vaccine targeting Globo H, a tumor-associated carbohydrate antigen expressed in many epithelial cancers. It is used in combination with OBI-821, an adjuvant designed to enhance the immune response. Previous studies have demonstrated that OBI-833/OBI-821 can elicit immune responses and provide disease stabilization in some cancer patients. Notably, Globo H expression has been detected in about 41% of intrahepatic cholangiocarcinoma specimens, providing a rationale for investigating this approach in biliary tract cancer.

The study design involves enrolling 30 patients in a single-arm trial. Eligible patients must have Globo H-positive advanced biliary tract cancer that has not progressed after 3±1 months of first-line gemcitabine/cisplatin therapy. Patients will receive OBI-833/OBI-821 subcutaneously on a gradually decreasing frequency schedule for up to 80 weeks, while continuing their gemcitabine/cisplatin regimen. The primary endpoint of the study is progression-free survival, with secondary endpoints including overall survival, tumor response, safety, and correlations between Globo H expression/antibodies and survival outcomes.

To ensure safety, the study incorporates a lead-in safety cohort of 6 patients before proceeding to full enrollment. Following the treatment period, patients will be followed for survival for up to 12 months after the end of treatment. This single-arm design allows for an efficient assessment of efficacy signals that could inform potential further development of this therapeutic approach.

The overall aim of the study is to evaluate whether adding OBI-833/OBI-821 maintenance therapy can prolong disease control in this patient population with high unmet medical need. By focusing on patients with Globo H-positive tumors who have initially responded to standard chemotherapy, the study seeks to explore a potentially targeted approach to maintaining and extending the benefits of first-line treatment in advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 20 years.
2. Histologically confirmed, unresectable advanced or metastatic biliary tract cancer, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma.
3. Patient with previously untreated disease if unresectable or metastatic at initial diagnosis will be eligible.
4. Patient with recurrent disease >6 months after curative surgery or >6 months after the completion of adjuvant therapy (chemotherapy and/or radiation) will be eligible.
5. Patient must have a documented Globo H H-score of at least 80 using a validated central IHC assay.
6. Patient must have received 3±1 months of the first-line GemCis regimen (gemcitabine, 1000 mg/m2 and cisplatin, 25 mg/m2 on days 1 and 8 of each 21-day cycle), have achieved SD, PR, or CR before enrollment (as confirmed by the Investigator), and plan to continue the GemCis regimen.
7. At least one measurable tumor lesion according to RECIST version 1.1 as assessed by the Investigator (local radiological image assessment).
8. Life expectancy ≥ 6 months.
9. East Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Organ function requirements - Subjects must have adequate organ functions as defined below:

    AST/ALT ≤ 3X ULN (upper limit of normal); AST/ALT ≤ 5X ULN in the presence of liver metastases Total bilirubin ≤ 2.0 X ULN Serum creatinine ≤ 1.5X ULN ANC ≥ 1,5500 /µL Platelets ≥ 100,000/µL
11. All eligible patients of childbearing potential must use effective contraception during study treatment, and for at least 2 months after the last dose of OBI-833/OBI-821. Subjects not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in the study. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
12. Understand and provide a written informed consent document according to institutional guidelines.

Exclusion Criteria:

1. Patient who has CNS metastasis or spinal cord compression.
2. Patient who is pregnant or breast-feeding at entry.
3. Patient with splenectomy.
4. Patient with HIV infection, active hepatitis B infection, or active hepatitis C infection. Patients with hepatitis B infection under anti-HBV medications are exceptionalcan be included in the study. Patients with hepatitis C infection history but inactive status are exceptionalcan be included in the study.
5. Patient with any autoimmune or other disorders requiring IV/oral steroids or immunosuppressive or immunomodulatory therapies.

   (e.g., type 1 juvenile onset diabetes mellitus, antibody positive for rheumatoid arthritis, Graves disease, Hashimoto thyroiditis, lupus, scleroderma, systemic vasculitis, hemolytic anemia, immune mediated thrombocytopenia, Crohn disease, ulcerative colitis, and psoriasis).
6. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0), except for alopecia and laboratory values listed in the inclusion criteria.
7. A history of other malignancies (except non-melanoma skin carcinoma, carcinoma in situ of the uterine cervix, follicular or papillary thyroid cancer) within 5 years.
8. Patient with any known uncontrolled comorbid illness including ongoing or active infections, symptomatic congestive heart failure (NYHA>2), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Treatment with any of the following therapies within 4 weeks prior to the first dose of OBI-833/OBI-821:

   * Anti-cancer therapies, including chemotherapy and targeted therapy (except the GemCis regimen).
   * Radiotherapy.
   * Immunotherapy, including monoclonal antibodies, cytokines, interferons, and checkpoint inhibitors.
   * Immunosuppressants, including cyclosporin, rapamycin, tacrolimus, rituximab, alemtuzumab, natalizumab, and cyclophosphamide.
   * Other biologics, including G-CSF and other hematopoietic growth factors.
   * Live attenuated vaccines.
   * IV/oral steroids except single prophylactic use in CT/MRI scan or other one-time use in approved indications. Use of inhaled and topical (except on the injection site) steroids is allowed.
   * Alternative and complementary medicine that may affect the immune system.
   * Other investigational drugs.
10. Patient with any known severe allergies (e.g., anaphylaxis) to any active or inactive ingredients in the study drugs.
11. Any other reason that the investigator deems the patient to be unsuitable for the study.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 12 to 18 months of subject recruitment, 80 weeks of OBI-833/OBI-821 treatment, and another 1 year for overall survival follow-up.
  The time from start of treatment until disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | 12 to 18 months of subject recruitment, 80 weeks of OBI-833/OBI-821 treatment, and another 1 year for overall survival follow-up.
  The time from start of treatment until death from any cause
Best overall tumor response | 12 to 18 months of subject recruitment, 80 weeks of OBI-833/OBI-821 treatment, and another 1 year for overall survival follow-up.
  by RECIST 1.1 criteria
Adverse events | 12 to 18 months of subject recruitment, 80 weeks of OBI-833/OBI-821 treatment, and another 1 year for overall survival follow-up.
  Incidences of adverse events and serious adverse events, Local injection site reaction, Changes in laboratory tests, including hematology and serum chemistry, Changes in vital signs, Changes in physical examination
Correlation between anti-Globo H IgM and IgG concentrations and survival | 12 to 18 months of subject recruitment, 80 weeks of OBI-833/OBI-821 treatment, and another 1 year for overall survival follow-up.
  biomarker response and survival correlation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Nan Yeh, Principal Investigator — Department of Surgery, Chang Gung Memorial Hospital, Linkou, Taiwan
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
  - Chang-Gung Memorial Hospital, Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No